CLINICAL TRIAL: NCT02530541
Title: Pilot Trial Assessment of the Antimicrobial Efficacy of Medline 2% CHG Cloth Preoperative Skin Preparation
Brief Title: Antimicrobial Efficacy of 2% CHG (Chlorhexidine Gluconate)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R14-015
Record Dates: First submitted 2015-08-16; First posted 2015-08-21 (Estimated); Results first posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2020-09

CONDITIONS: Healthy
MeSH Terms: interventions — chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CHG 1 min (Experimental): 1 min application time
  Interventions: Drug: CHG
- CHG 2 min (Experimental): 2 min application time
  Interventions: Drug: CHG
- Comparator CHG (Active Comparator): Marketed CHG
  Interventions: Drug: CHG

INTERVENTIONS:
Drug: CHG — Varied application times
  Other Names: Chlorhexidine Gluconate

SUMMARY:
Pilot study to evaluate and compare activity of preoperative preparation with comparator

DETAILED DESCRIPTION:
Evaluate and compare similar preoperative surgical preparations in healthy volunteers. Various application times were evaluated. Efficacy was assess using TFM criteria.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* No dermatological conditions

Exclusion Criteria:

* Sensitivity to CHG
* Sensitivity to natural latex rubber or adhesive skin products

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Campbell, Principal Investigator — Bioscience Labs

IPD SHARING:
Plan to Share IPD: Yes
Data to be shared with FDA

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Upon achieving sufficient microbial growth prior to product application on either the abdomen, groin or both abdomen and groin regions, sites of the participant were then randomized to receive one or two products for evaluation for up to 4 sites. Differences in the number of participants is based on microbial qualifications.
Pre-assignment Details: Participants were randomized to be treated with at least 2 treatments/ Arms (out of 3) at the same time for both groin and abdomen. Total numbers represent sites not the individual number of participants.
Units Other Than Participants: sites
Groups:
- CHG 1 Min Abdomen: CHG 1 min Abdomen sites
- CHG 2 Min Abdomen: CHG 2 min Abdomen sites
- Comparator CHG Abdomen; Comparator CHG Groin: Marketed CHG - only applied per products instructions for use
- CHG 1 Min Groin: CHG 1 min Groin sites
- CHG 2 Min Groin: CHG 2 min Groin sites
Period: Overall Study
Arm/Group | CHG 1 Min Abdomen | CHG 2 Min Abdomen | Comparator CHG Abdomen | CHG 1 Min Groin | CHG 2 Min Groin | Comparator CHG Groin
Started | 21; 21 sites | 23; 23 sites | 22; 22 sites | 21; 21 sites | 20; 20 sites | 19; 19 sites
Completed (33 were treated with both interventions, though interventions differ with application time. 24 subjects completed with passing treatment baseline values) | 14; 14 sites | 15; 15 sites | 14; 14 sites | 15; 15 sites | 15; 15 sites | 14; 14 sites
Not Completed | 7; 7 sites | 8; 8 sites | 8; 8 sites | 6; 6 sites | 5; 5 sites | 5; 5 sites

BASELINE CHARACTERISTICS:
Population: Participants received up to 2 treatments at the same time. The treatments included 2 different testing sites.
Groups:
- CHG 1, CHG 2, Comparator CHG: Participants could receive up to 2 different treatments at the same time. Treatments included CHG at 1 min, CHG at 2 min or Comparator CHG.
Arm/Group | CHG 1, CHG 2, Comparator CHG
Number analyzed (Participants) | 33
Age, Customized [Mean (Full Range); unit: years]
  Age | 48 [19 to 79]
Sex: Female, Male [Count of Participants; unit: Participants] — 33 participants were evaluated with up to 2 products. However only participants that achieved baseline criteria based on post testing analysis were used in the final analysis. The total of participants used was 21.
  Participants
    Female | 21
    Male | 12
Region of Enrollment [Number; unit: Sites exposed]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Log Reduction of Bacterial Flora on the Abdomen and Groin
Description: Evaluate the Log Reduction of normal flora at various timepoints.
Time Frame: 10 min, 6 hr and 8 hr
Population: Determine 70% responder rates
Measure: Mean (Standard Deviation); unit: Log10 Reductions
Units Other Than Participants: Sites Exposed
Groups:
- CHG 1 Min Abdomen; CHG 1 Min Groin: 1 min application time
- CHG 2 Min Abdomen; CHG 2 Min Groin: 2 min application time
- Comparator CHG Abdomen: Marketed CHG Standard Application Time
- Comparator CHG Groin: Comparator CHG Standard Application Time
Arm/Group | CHG 1 Min Abdomen | CHG 2 Min Abdomen | Comparator CHG Abdomen | CHG 1 Min Groin | CHG 2 Min Groin | Comparator CHG Groin
Number analyzed (Participants) | 21 | 23 | 22 | 21 | 20 | 19
Number analyzed (Sites Exposed) | 21 | 23 | 22 | 21 | 20 | 19
Log10 Reductions
  10 min | 1.9 (1.6) | 2.0 (1.5) | 1.3 (1.8) | 1.9 (0.6) | 2.4 (1.1) | 2.1 (1.1)
  6 hour | 2.6 (1.3) | 2.5 (1.4) | 1.7 (1.6) | 2.3 (0.8) | 2.8 (1.2) | 1.9 (0.8)
  8 hour | 2.6 (1.0) | 2.2 (1.6) | 1.4 (1.2) | 2.5 (0.9) | 2.7 (0.8) | 2.2 (1.1)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from baseline out to 8 hours.
Description: Participants received up to 2 products at the same time.
Groups:
- CHG 1 Min, CHG 2 Min, Comparator CHG: 1 min application time, 2 min application time or comparator application. Up to 2 products applied to the same participant.
Arm/Group | CHG 1 Min, CHG 2 Min, Comparator CHG
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 0/33

LIMITATIONS AND CAVEATS:
Small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data considered confidential